CLINICAL TRIAL: NCT06824480
Title: The Effect of Debriefing of Childbirth in the Early Postpartum Period on the Psychological Outcomes
Brief Title: The Effect of Postpartum Debriefing on the Psychological Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gozde Gokce Isbir, PROFESSOR, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VBalci
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-02

CONDITIONS: Well-Being, Psychological
Keywords: debriefing, trauma, fear, depression
MeSH Terms: conditions — Psychological Well-Being; Wounds and Injuries; Depression | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental: debriefing grup (Experimental): Women who volunteered to participate in the study and met the participation criteria were informed about the study. The first session will be held face to face in the clinic for 40 minutes. Then, the second session will be held by phone within 4-6 weeks after birth, with a total of 2 meetings with each woman for approximately 40 minutes.
  Interventions: Behavioral: debriefing group
- experimental: control grup (Experimental): The women in the control group will be asked how the birth went within 12-24 hours after birth by the researcher as part of their routine care, but no detailed analysis or interpretation will be made.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: debriefing group — Women who volunteered to participate in the study and met the participation criteria were informed about the study. The first session will be held face to face in the clinic for 40 minutes. Then, the second session will be held by phone within 4-6 weeks after birth, with a total of 2 meetings with each woman for approximately 40 minutes.
  Arms: experimental: debriefing grup
Behavioral: control group — he women in the control group will be asked how the birth went within 12-24 hours after birth by the researcher as part of their routine care, but no detailed analysis or interpretation will be made.
  Arms: experimental: control grup

SUMMARY:
This study was planned to determine the effect of re-signification of birth in the early postpartum period on postpartum fear of childbirth, postpartum depression and birth trauma.

DETAILED DESCRIPTION:
This study was contucted between february 2024 and June 2025 in Turkey , as a single-blind randomized controlled experimental study to determine the effect of reinterpretation of birth on postpartum fear of childbirth, postpartum depression and birth trauma.During data collection, participants were informed about the purpose of the study and those who volunteered to participate in the research were accepted into the study by signing an informed consent form.Data; When the study was approved, it was planned to be collected face to face within the first 12-24 hours after birth and by telephone within 6-8 weeks after birth. CONSORT directive was followed in the research planning.

ELIGIBILITY:
Inclusion Criteria:

Women who volunteer to participate in the study, Whose mother tongue is Turkish, Who are between the ages of 18-45, Who are at least primary school graduates, Who are 37-42 weeks pregnant, Who are nulliparous, Who have a healthy pregnancy, Who do not have a psychological condition or psychiatric disorder, Who are monitored and cared for in the first 24 hours after birth at the Tarsus State Hospital Maternity Department, Who approve of the reinterpretation of birth application to be carried out by the researcher will be included in the sample.

Exclusion Criteria:

Those who did not volunteer to participate in the study, Those who gave birth before the 37th week of pregnancy, Those who were multiparous, Those who had abnormal medical conditions during pregnancy (placental disorder, preeclampsia, premature birth threat, etc.),

Those whose native language is not Turkish, Those who have visual, speech and hearing impairments, Those who had an emergency cesarean section, Those who stayed in the hospital for less than 12 hours after birth, Those who received a psychiatric diagnosis during the postpartum period (except those diagnosed with postpartum depression and post-traumatic stress disorder related to birth), Those who could not be reached by phone during the follow-up of the study, Women who developed complications in the first 24 hours after birth and required intensive care, Those whose babies required neonatal intensive care during the postpartum period, Those who experienced another life event that traumatized the woman during the postpartum period (harassment, rape, earthquake, accident, loss of a loved one) etc.) Those who want to withdraw from the study at any stage of the study will not be included in the sample.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 72 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | the first 12-24 hours after birth
  It includes women's sociodemographic characteristics, education and employment status, and contact information.
Birth Process Evaluation Form | the first 12-24 hours after birth
  It consists of 22 questions that include obstetric characteristics related to labor (gestational week, pregnancy planning/desire) and interventions performed during birth.
Wijma Birth Expectation/Experience Scale B version (W-DBÖ-B) at Birth: | the first 12-24 hours after birth
  Wijma Birth Expectation/Experience Scale (W-DEQ) was developed by Klaas and Barbro Wijma (1998) to measure the fear of birth experienced by women. The scale consists of 32 items. The answers on the scale are numbered from 0 to 5 and are in the six-point Likert type. 0 is expressed as "completely" and 5 is expressed as "not at all". The minimum score on the scale is 0, while the maximum score is 160. As the score increases, the fear of childbirth experienced by women increases. Questions numbered 2, 3, 6, 7, 10, 11, 14, 18, 19, 23, 24, 26, 30 are calculated by reversing the scale. The scale, which was adapted to Turkish by Körükcü, Bulut and Kukulu and its validity and reliability were made, has six sub-dimensions. These dimensions are determined as Anxiety about contractions (items 1,2,6,11,15,16,18,23), inadequacy in positive behaviors (items 24,25,26,30), loneliness (items 3,7,10,14,19,21,22
Wijma Birth Expectation/Experience Scale B version (W-DBÖ-B) at Birth: (ANNEX-3) | first 6-8 weeks after birth
  Wijma Birth Expectation/Experience Scale (W-DEQ) was developed by Klaas and Barbro Wijma (1998) to measure the fear of birth experienced by women. The scale consists of 32 items. The answers on the scale are numbered from 0 to 5 and are in the six-point Likert type. 0 is expressed as "completely" and 5 is expressed as "not at all". The minimum score on the scale is 0, while the maximum score is 160. As the score increases, the fear of childbirth experienced by women increases. Questions numbered 2, 3, 6, 7, 10, 11, 14, 18, 19, 23, 24, 26, 30 are calculated by reversing the scale. The scale, which was adapted to Turkish by Körükcü, Bulut and Kukulu and its validity and reliability were made, has six sub-dimensions. These dimensions are determined as Anxiety about contractions (items 1,2,6,11,15,16,18,23), inadequacy in positive behaviors (items 24,25,26,30), loneliness (items 3,7,10,14,19,21,22
City Birth Trauma Scale (CityBiTS) | first 6-8 weeks after birth
  The City Birth Trauma Scale (CityBiTS) was developed by Susan Ayers and colleagues to assess PTSD and its symptoms in the postpartum period. The original measurement tool had a Cronbach's Alpha coefficient of 0.92 for the entire scale and between 0.82 and 0.88 for the subscales The scale consists of 29 items and is a four-point Likert-type scale. The scale assesses symptoms of stress (items 1-2), re-experiencing (items 3-7), avoidance (items 8-9), negative cognitions and mood (items 10-16), and hyperarousal (items 17-22). In addition, items 23 and 24 of the scale focus on dissociative symptoms, with a score of "0" in item 25 indicating pre-partum onset of PTSD and a score of "2" indicating delayed onset PTSD. The duration of symptoms is assessed with item 26. While distress and impairment symptoms are assessed with items 27 and 28, the last item of the scale (item 29) is the exclusion criterion for PTSD . Items 3-22 can be scored on the scale and a score between 0-60 can be.
Edinburgh Postpartum Depression Scale (EDPS) | first 6-8 weeks after birth
  EPDS was developed by Cox and colleagues in 1987 and is a measurement tool that determines the risk, level, and severity of depression in the postpartum period. The scale is a self-assessment scale. The measurement tool consists of 10 items on a four-point Likert-type scale evaluated between 0 and 3. The highest score that can be obtained from the scale is 30. Questions 1, 2, and 4 on the scale are scored in the format 0-1-2-3, while questions 3, 5, 6, 7, 8, 9, and 10 are scored in the format 3-2-1-0. The cut-off point of the scale was calculated as 13. Cronbach's alpha value of the original version of EPDS was determined as 0.87. The Turkish validity and reliability study of the scale was conducted by Aydın and his colleagues in 2004, and Cronbach's alpha value was determined as 0.72.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Mersin university, Mersin
  - Mersin University, Mersin

IPD SHARING:
Plan to Share IPD: No